CLINICAL TRIAL: NCT04525937
Title: Racial and Economic Disparities and Unmet Needs in Patients With Severe Aortic Valvular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Racial Disparities
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Disparities in Treatment of Aortic Valve Stenosis; Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Disparities
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Severe Aortic Stenosis with Disparities: Patients will complete a survey and their aortic stenosis will be clinically followed at 30 days and one year
  Interventions: Other: Patient Questionnaire
- Medical Providers with Disparities: Referring primary care providers complete a questionnaire on their referral practices for patients with severe aortic stenosis
  Interventions: Other: Provider Questionnaire

INTERVENTIONS:
Other: Patient Questionnaire — Patient Questionnaire
  Groups: Patients with Severe Aortic Stenosis with Disparities
Other: Provider Questionnaire — Provider Questionnaire
  Groups: Medical Providers with Disparities

SUMMARY:
Common barriers to receiving appropriate guideline-driven care for patients with severe aortic stenosis include referral biases by primary care providers (lack of provider education), patient comorbidities (degree of fragility), as well as psychosocial issues and cultural barriers. Additionally, race, ethnicity, socioeconomic status (SES) and education level are shown to be persistent barriers to accessing healthcare services and healthcare systems, creating a significant practice gap between various patient populations. The most recent transcatheter valve therapies (TVT) registry data show that >94% of TAVR recipients are Caucasian, followed by less than 4% of African-Americans and Hispanics, respectively. There is a critical need to understand the barriers to treatment and care among severe aortic valve disease patients of disparate groups. This study is a multi-center, retrospective and prospective cohort study of patients diagnosed with severe aortic stenosis. Additionally, we will be surveying referring primary care providers, cardiologists and cardiovascular surgeons to assess their current referral practices for patients with severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Disparity/Diversity background (either race/ethnicity, low SES (adults with incomes at or below the federal poverty level (family income to poverty ratio, ≤1), language (non-English speaker) or education (≤9 years of education))
* Patient scheduled for transcatheter aortic valve replacement using the Edwards Sapien valve, OR recently implanted with Edwards Sapien valve (up to 1 year post-TAVR)
* Echocardiographic diagnosis of severe, symptomatic AS and intermediate to high surgical risk per Society of Thoracic Surgeons (STS) mortality risk-score

Exclusion Criteria:

* Age < 18
* Patients who do not allow their records to be used for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients:
  - Over 18 years of age with echocardiographic diagnosis of severe, symptomatic AS and intermediate to high surgical risk per Society of Thoracic Surgeons (STS) mortality risk-score who have a disparate condition
  Providers:
  - Referring primary care providers, cardiologists and cardiovascular surgeons at the study sites.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient Mortality | 30 days and 1 year
MACE (Major Adverse Cardiac Event) | 30 days and 1 year

SECONDARY OUTCOMES:
Referring physician- related barriers/biases. | through study completion, an average of 1 year
  Secondary outcomes (Providers): referring physician-related barriers/biases against routine guideline-driven care for members of disparate groups with severe aortic stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Goessl, MD, PhD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No